CLINICAL TRIAL: NCT02205593
Title: A Prospective, Randomized, Controlled Study of the Impact of Education and Stress-reduction Techniques on Psoriasis and Eczema.
Brief Title: Haut-Tief Patient Education on Psoriasis and Eczema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Haut-Tief
Record Dates: First submitted 2014-07-14; First posted 2014-07-31 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis; Atopic Dermatitis/ Eczema
Keywords: psoriasis; atopic dermatitis; eczema; patient education; stress reduction; quality of life
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): patient group receiving regular follow-up visits (baseline, 3 months, 6 months, 9 months)
  Interventions: Behavioral: Control
- Haut Tief patient education (Active Comparator): patient group receives the educational program with regular follow-up visits (baseline, 3 months, 6 months, 9 months).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Regular follow-up and treatment WITHOUT behavioural intervention

SUMMARY:
'Haut-Tief' (Skin Deep) is an educational, stress reducing program for patients with psoriasis or atopic dermatitis. A range of support activities will be offered in order to learn effective self-management strategies and attitude to one's chronic skin disease and consequently improving quality of life.

DETAILED DESCRIPTION:
The educational program consists of 2-hours of educational (dermatology, specialized nurse, psychologist) and stress-reduction sessions (yoga, meditation, physiotherapy) twice a week during 9 weeks.

A multidisciplinary team of trainers is involved. Primary endpoint is the general and skin dependent quality of life measured by questionnaires. HRQoL (Health-Related Quality of Life) is measured at baseline, after 3 months, 6 months and 9 months follow up. Patients are recruited from the out-patient clinic at the Department of Dermatology of the University Hospital Zurich. Patients are randomized in an intervention and control group. Intervention group receives the education program additionally to follow-up visits whereas the control group receives follow-up visits. Several runs are planned.

ELIGIBILITY:
Inclusion Criteria:

* Chronic psoriasis (disease for more than 3 months)
* Chronic eczema (disease for more than 3) months)
* Age ≥ 18 years
* Oral and written informed consent

Exclusion Criteria:

* systemic antiinflammatory therapy
* treatment with other investigational products
* other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc),
* known or suspected non-compliance, drug or alcohol abuse,
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject
* participation in another study within the 30 days preceding and during the present study, (viii) previous enrollment into the current study,
* enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
change in DLQI (Dermatology Life Quality Index) score [ ] | baseline, 3 months, 6 months, 9 months
  DLQI is a questionnaire measuring Health related quality of life 10 questions
change in Skindex-29 score [ ] | baseline, 3 months, 6 months, 9 months
  Questionnaire measuring Health related quality of life 29 questions
change in ShortForm 36 score [ ] | baseline, 3 months, 6 months, 9 months
  Questionnaire measuring Health related quality of life
change in EQ 5D score [ ] | baseline, 3 months, 6 months, 9 months
  Questionnaire measuring Health related quality of life
change in EQ VAS (EQ visual analogue scale) score [ ] | baseline, 3 months, 6 months, 9 months
  Questionnaire measuring Health related quality of life

SECONDARY OUTCOMES:
change in EASI (eczema area and severity index) score [ ] | baseline, 3 months, 6 months, 9 months
  clinical score for atopic dermatitis
change in PASI (psoriasis area and severity index) [ ] | baseline, 3 months, 6 months, 9 months
  clinical score for psoriasis
BDI (Beck Depression Inventory) score [ ] | baseline, 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Hofbauer, Prof MD, Principal Investigator — University Hospital Zurich, Dept. of Dermatology
Locations (1):
- University Hospital Zurich, Department of Dermatology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No